CLINICAL TRIAL: NCT03326154
Title: Health Related Quality of Life and Abdominal Symptoms After Cholecystectomy
Brief Title: Post-Cholecystectomy Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hanna Lampela, Ph.D., Helsinki University Central Hospital
Other Study IDs: HUS/2317/2016
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Gallstone
Keywords: cholecystectomy; quality of life
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, observational — Observation

SUMMARY:
The study aims to identify factors associated with no increase in gastrointestinal quality of life after elective cholecystectomy for gallstones.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic cholecystectomy patients
* indication for operation symptomatic gallstones

Exclusion Criteria:

* previous complication of gallstone disease
* indication for cholecystectomy other than symptomatic gallstones
* illness significantly lowering quality of life
* inability to fill in questionnaires
* denies participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life: Gastrointestinal Quality of Life GIQLI score | 1 year
  10 point improvement in Gastrointestinal Quality of Life GIQLI score

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Lampela, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Jorvi, Helsinki University Hospital, Espoo
  - HUS Hyvinkää Hospital, Hyvinkää